CLINICAL TRIAL: NCT02102464
Title: Pilot Study for Treatment of Meibomian Gland Dysfunction and Evaporative Dry Eye in Contact Lens Wearers
Brief Title: Treatment of Meibomian Gland Dysfunction and Dry Eye in Contact Lens Wearers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TearScience, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LF006
Record Dates: First submitted 2014-03-30; First posted 2014-04-03 (Estimated); Results first posted 2017-09-18 (Actual); Last update posted 2017-10-18 (Actual); Status verified 2017-09

CONDITIONS: Meibomian Gland Dysfunction; Dry Eye
MeSH Terms: conditions — Meibomian Gland Dysfunction; Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- LipiFlow (Experimental): Single 12-minute LipiFlow treatment
  Interventions: Device: LipiFlow treatment
- Untreated Control (No Intervention): Untreated Control (No Intervention)
- Crossover LipiFlow Treatment (Experimental): Crossover LipiFlow treatment of the untreated control group after 3 months
  Interventions: Device: LipiFlow treatment

INTERVENTIONS:
Device: LipiFlow treatment — The LipiFlow® Thermal Pulsation System is a prescription device intended for the application of localized heat and pressure therapy in adult patients with chronic cystic conditions of the eyelids, including meibomian gland dysfunction, also known as evaporative dry eye or lipid deficiency dry eye.
  Other Names: LipiFlow® Thermal Pulsation System
  Arms: Crossover LipiFlow Treatment; LipiFlow

SUMMARY:
The pilot study objective is to evaluate the potential benefits of LipiFlow® System treatment of contact lens wearers with meibomian gland dysfunction and evaporative dry eye by assessing for improvement in meibomian gland function and reduction of dry eye symptoms in comparison to an untreated control.

DETAILED DESCRIPTION:
This is a prospective, non-significant risk, open-label, randomized clinical trial of LipiFlow® treatment of contact lens wearers with meibomian gland dysfunction and evaporative dry eye. All subjects undergo examination to determine study eligibility and to capture the Baseline status. Subjects are randomized to receive LipiFlow® treatment (Treatment Group) or no LipiFlow® treatment (Untreated Control Group). The Treatment group is evaluated one month after receiving LipiFlow® treatment. Study endpoints are evaluated at 3 Months by comparing the Treatment Group to the Untreated Group. To facilitate subject recruitment, the Untreated Control group receives Crossover LipiFlow® treatment (Crossover Treatment Group) at 3 Months. The Crossover Treatment group is evaluated one month after receiving LipiFlow® treatment (4 Months visit).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of meibomian gland dysfunction and dry eye
* At least 18 years of age
* Willing to comply with randomization, attend all study visits and follow patient instructions
* Habitual soft contact lens wearer 2 to 18 hours/day and 4 to 7 days/week
* No change in contact lens type or dimensions for the past 3 months
* Clinician assessment of acceptable contact lens fit and disinfecting solution
* Tear film interferometry of 100 units or less

Exclusion Criteria:

* Systemic disease conditions that cause dry eye
* Use of systemic medications known to cause dryness
* History of any of the following ocular conditions in the past 3 months: surgery, trauma, Herpes infection, recurrent inflammation, punctal plug insertion or punctal occlusion
* Presence of any of the following active conditions: ocular infection, ocular inflammation, moderate to severe allergic conjunctivitis, severe eyelid inflammation, eyelid abnormality that affects lid function, or ocular surface abnormality that compromises corneal integrity
* Use of other treatments for meibomian gland dysfunction or dry eye except over the counter lubricants or dietary supplements
* Participation in another ophthalmic drug or device trial in the past month
* Employee, relative of employee or associate of the clinical site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2014-04; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christy Coleman, OD, MPH, Study Director — TearScience, Inc.
Locations (6):
- United States (5):
  - School of Optometry, The University of Alabama at Birmingham, Birmingham, Alabama
  - Clayton Eye Center, Morrow, Georgia
  - Charlotte Eye Ear Nose and Throat Associates, P.A., Charlotte, North Carolina
  - May Eye Care Center & Associates, Hanover, Pennsylvania
  - Specialty Eyecare Group, Kirkland, Washington
- Centre for Contact Lens Research, Waterloo, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Eyes
Groups:
- Crossover LipiFlow: Untreated Control Subjects received a 12-minute LipiFlow treatment after the 3-month visit
Period: Randomized Study
Arm/Group | LipiFlow | Untreated Control | Crossover LipiFlow
Started | 29; 58 Eyes | 26; 52 Eyes | 0; 0 Eyes
Completed | 29; 58 Eyes | 25; 50 Eyes | 0; 0 Eyes
Not Completed | 0; 0 Eyes | 1; 2 Eyes | 0; 0 Eyes
Not completed — Withdrawal by Subject | 0 | 1 | 0
Period: Crossover LipiFlow Treatment of Control
Arm/Group | LipiFlow | Untreated Control | Crossover LipiFlow
Started | 0; 0 Eyes | 0; 0 Eyes | 25; 50 Eyes
Completed | 0; 0 Eyes | 0; 0 Eyes | 25; 50 Eyes
Not Completed | 0; 0 Eyes | 0; 0 Eyes | 0; 0 Eyes

BASELINE CHARACTERISTICS:
Units Other Than Participants: Eyes
Groups:
- Total: Total of all reporting groups
Arm/Group | LipiFlow | Untreated Control | Total
Number analyzed (Participants) | 29 | 26 | 55
Number analyzed (Eyes) | 58 | 52 | 110
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.0 (13.1) | 43.5 (15.9) | 41.7 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 22 | 47
  Male | 4 | 4 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 29 | 25 | 54
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 6 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 4 | 9
  White | 17 | 16 | 33
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 8 | 8 | 16
  United States | 21 | 18 | 39
Meibomian Gland Score [Mean (Standard Deviation); unit: units on a scale] — Along the lower lid, secretion characteristics of 15 meibomian glands were evaluated including five glands each in the temporal, central and nasal regions of the lower eyelid. For each gland, secretion characteristics were graded as 3 (clear liquid), 2 (cloudy liquid), 1 (inspissated/ toothpaste consistency) and 0 (no secretion). The total meibomian gland score is the sum of the grades for all 15 glands with a range between 0 and 45. A higher score reflects less meibomian gland dysfunction.
  units on a scale | 8.0 (3.5) | 8.2 (4.2) | 8.1 (3.8)
SPEED Score [Mean (Standard Deviation); unit: units on a scale] — Using Standard Patient Evaluation of Eye Dryness (SPEED) questionnaire, symptoms evaluated were dryness, grittiness or scratchiness; soreness or irritation; burning or watering; and eye fatigue. Frequency scale: 0 (never), 1 (sometimes), 2 (often) and 3 (constant). Severity scale: 0 (no problems), 1 (tolerable-not perfect but not uncomfortable), 2 (uncomfortable-irritating but does not interfere with my day), 3 (bothersome-irritating and interferes with my day) and 4 (intolerable-unable to perform my daily tasks). SPEED score is the sum of frequency and severity scores (range 0 to 28).
  units on a scale | 14.5 (4.8) | 15.3 (4.5) | 14.9 (4.6)
Comfortable Contact Lens Wear Time [Mean (Standard Deviation); unit: hours per day] — Subjects reported how long they wore their contact lenses each day (total contact lens wear time), and how long the contact lens wear was comfortable (comfortable contact lens wear time).
  hours per day | 5.4 (3.4) | 4.3 (3.1) | 4.9 (3.3)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Meibomian Gland Score From Baseline at 3 Months
Description: The Primary Endpoint was intended to assess for improvement in meibomian gland function in symptomatic contact lens wearers after LipiFlow treatment in comparison to an untreated control.The Primary Endpoint was defined as the mean change in meibomian gland score in the LipiFlow Treatment group compared to Untreated Control group from Baseline to 3 Months. To determine the meibomian gland score, secretion characteristics of 15 meibomian glands along the lower eyelid were evaluated including five glands each in the temporal, central and nasal regions of the lower eyelid. For each gland, secretion characteristics were graded as 3 (clear liquid), 2 (cloudy liquid), 1 (inspissated/ toothpaste consistency) and 0 (no secretion). The total meibomian gland score is the sum of the grades for all 15 glands with a range between 0 and 45. A higher score reflects less meibomian gland dysfunction.
Time Frame: 3 Months
Population: Intent to Treat (ITT) Population of all randomized subjects.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | LipiFlow | Untreated Control
Number analyzed (Participants) | 29 | 25
Number analyzed (Eyes) | 58 | 50
units on a scale | 12.4 [10.0 to 14.8] | 1.4 [-0.4 to 3.3]
Statistical Analysis 1: Comparison: LipiFlow vs Untreated Control; Test type: Superiority; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = 11.0, 95% CI 2-sided [8.0 to 14.0]

2. Secondary Outcome: Mean Change in Dry Eye Questionnaire Score From Baseline at 3 Months
Description: The Secondary Endpoint was intended to assess for reduction in dry eye symptoms in symptomatic contact lens after LipiFlow treatment in comparison to an untreated control using the Standard Patient Evaluation of Eye Dryness (SPEED) questionnaire. The Secondary Endpoint was defined as the mean change in SPEED score in the LipiFlow Treatment group compared to Untreated Control group from Baseline to 3 Months. Dry eye symptoms evaluated were dryness, grittiness or scratchiness; soreness or irritation; burning or watering; and eye fatigue. Symptom frequency and severity were assessed. The SPEED score is the sum of frequency and severity scores with a range from 0 to 28. A lower SPEED score represents less frequent and/or less severe symptoms.
Time Frame: 3 Months
Population: Intent to Treat (ITT) Population of all randomized subjects.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | LipiFlow | Untreated Control
Number analyzed (Participants) | 29 | 25
units on a scale | -8.4 [-10.2 to -6.6] | -0.7 [-2.5 to 1.1]
Statistical Analysis 1: Comparison: LipiFlow vs Untreated Control; Test type: Superiority; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = -7.7, 95% CI 2-sided [-10.2 to -5.2]

3. Other Pre Specified Outcome: Mean Change in Comfortable Contact Lens Wear Time From Baseline at 3 Months
Description: Subjects reported how long they wore their contact lenses per day (total contact lens wear time) and how long the contact lenses were comfortable (comfortable contact lens wear time). A pre-specified exploratory analysis was to compare the mean change in comfortable contact lens wear time between Baseline and 3 Months for the LipiFlow group vs. untreated control.
Time Frame: 3 Months
Population: Intent to Treat (ITT) of all randomized subjects
Measure: Mean (95% Confidence Interval); unit: hours per day
Arm/Group | LipiFlow | Untreated Control
Number analyzed (Participants) | 29 | 25
hours per day | 3.7 [2.8 to 4.5] | -0.3 [-0.8 to 0.3]
Statistical Analysis 1: Comparison: LipiFlow vs Untreated Control; Test type: Superiority; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = 3.9, 95% CI 2-sided [2.5 to 5.4]

4. Other Pre Specified Outcome: Mean Change in Meibomian Gland Score From Baseline at 1 Month
Description: The mean change in meibomian gland score from Baseline was also evaluated at 1 Month post-LipiFlow treatment for the LipiFlow and Crossover LipiFlow Groups. The LipiFlow Group was assessed at the 1-Month visit. The Crossover LipiFlow Group was assessed at the 4-Month visit (one month after receiving crossover LipiFlow treatment). There was no planned statistical analysis comparison between the LipiFlow and Crossover LipiFlow groups at 1 Month. To determine the meibomian gland score, secretion characteristics of 15 meibomian glands along the lower eyelid were evaluated including five glands each in the temporal, central and nasal regions of the lower eyelid. For each gland, secretion characteristics were graded as 3 (clear liquid), 2 (cloudy liquid), 1 (inspissated/ toothpaste consistency) and 0 (no secretion). The total meibomian gland score is the sum of the grades for all 15 glands with a range between 0 and 45. A higher score reflects less meibomian gland dysfunction.
Time Frame: 1 Month
Population: Intent to Treat (All randomized subjects)
Measure: Mean (95% Confidence Interval); unit: units on a scale
Units Other Than Participants: Eyes
Groups:
- Crossover LipiFlow Group: Untreated Control Subjects received a 12-minute LipiFlow treatment after the 3-month visit
Arm/Group | LipiFlow | Crossover LipiFlow Group
Number analyzed (Participants) | 29 | 25
Number analyzed (Eyes) | 58 | 50
units on a scale | 11.7 [9.2 to 14.2] | 14.3 [11.1 to 17.5]

5. Other Pre Specified Outcome: Mean Change in Dry Eye Questionnaire From Baseline at 1 Month
Description: The mean change in dry eye symptoms from Baseline based on the SPEED questionnaire score was also evaluated at 1 Month post-LipiFlow treatment for the LipiFlow and Crossover LipiFlow Groups. The LipiFlow Group was assessed at the 1-Month visit. The Crossover LipiFlow Group was assessed at the 4-Month visit (one month after receiving cossover LipiFlow treatment). There was no planned statistical analysis comparison between the LipiFlow and Crossover LipiFlow groups at 1 Month. Dry eye symptoms evaluated were dryness, grittiness or scratchiness; soreness or irritation; burning or watering; and eye fatigue. Symptom frequency and severity were assessed. The SPEED score is the sum of frequency and severity scores with a range from 0 to 28. A lower SPEED score represents less frequent and/or less severe symptoms.
Time Frame: 1 Month
Population: Intent to Treat (All randomized subjects)
Measure: Mean (95% Confidence Interval); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | LipiFlow | Crossover LipiFlow
Number analyzed (Participants) | 29 | 25
Number analyzed (Eyes) | 58 | 50
units on a scale | -8.3 [-10.1 to -6.5] | -8.1 [-10.7 to -5.5]

6. Other Pre Specified Outcome: Mean Change in Comfortable Contact Lens Wear Time From Baseline at 1 Month
Description: Subjects reported how long they wore their contact lenses per day (total contact lens wear time) and how long the contact lenses were comfortable (comfortable contact lens wear time). The mean change in comfortable contact lens wear time from Baseline was also evaluated at 1 Month post-LipiFlow treatment for the LipiFlow and Crossover LipiFlow Groups. The LipiFlow Group was assessed at the 1-Month visit. The Crossover LipiFlow Group was assessed at the 4-Month visit (one month after receiving cossover LipiFlow treatment). There was no planned statistical analysis comparison between the LipiFlow and Crossover LipiFlow groups at 1 Month.
Time Frame: 1 Month
Population: Intent to Treat (all randomized subjects)
Measure: Mean (95% Confidence Interval); unit: hours per day
Units Other Than Participants: Eyes
Arm/Group | LipiFlow | Crossover LipiFlow Group
Number analyzed (Participants) | 29 | 25
Number analyzed (Eyes) | 58 | 50
hours per day | 4.0 [2.9 to 5.1] | 3.7 [2.5 to 4.8]

ADVERSE EVENTS:
Time Frame: Device-related adverse event data were analyzed over the entire study duration. For the LipiFlow Group, this time frame was 3 months. For the Crossover LipiFlow Group, the time frame was one month follow-up after receiving crossover LipiFlow treatment of the untreated control subjects at the 3-Month visit.
Description: An adverse event was defined as any untoward medical occurrence in a subject in association with use of the device or study procedure. Investigators were required to document adverse events and assess the causal relationship with the device or study procedure. The Medical Monitor reviewed adverse events as they were reported by Investigators.
Groups:
- Crossover LipiFlow Group: Untreated Control Group received a single 12-minute Crossover LipiFlow treatment at the 3-Months visit.
Arm/Group | LipiFlow | Untreated Control | Crossover LipiFlow Group
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/26 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/26 | 0/25
Other Adverse Events (participants affected / at risk) | 0/29 | 0/26 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Within 18 months of Sponsor's receipt of data from all sites, Investigators may publish or present the Investigator's individual results. Investigator must submit materials to Sponsor for review and comment at least 30 days prior to presentation or submission for publication. Investigator will consider all reasonable comments from Sponsor. Upon Sponsor's written request, Investigator agrees to delete any Proprietary Information other than Investigator's individual Study results.